CLINICAL TRIAL: NCT06321068
Title: Phase II/III Study of the Safety and Efficacy of BAT1308 in Combination With Platinum-containing Chemotherapy for First-line Treatment of Advanced or Recurrent Mismatch Repair Protein-deficient (dMMR) Endometrial Cancer
Brief Title: BAT1308 in Combination With Platinum-containing Chemotherapy is Used for the First-line Treatment of Advanced or Recurrent dMMR Endometrial Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the adjustment of our company's research and development strategy, we are now prematurely terminating this project.
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-1308-003-CR
Record Dates: First submitted 2024-01-07; First posted 2024-03-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAT1308 (Experimental): Strength 100 mg/4 mL, intravenous drip, recommended dose 300 mg, administered every 3 weeks (21 days) (Q3W)
  Interventions: Drug: carboplatin; Drug: Paclitaxel; Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection

INTERVENTIONS:
Drug: carboplatin — the usage and dosage should be determined by the investigator
  Other Names: Bobei
Drug: Paclitaxel — the usage and dosage should be determined by the investigator
  Other Names: Tesu
Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection — Strength 100 mg/4 mL, intravenous drip, recommended dose 300 mg, administered every 3 weeks (21 days) (Q3W).
  Other Names: BAT1308 injection

SUMMARY:
Phase II study: Safety and preliminary efficacy of BAT1308 combined with platinum-containing chemotherapy;Phase III study: Confirmatory safety and efficacy study of BAT1308 combined with platinum-containing chemotherapy for first-line treatment of advanced or recurrent mismatch repair protein-deficient (dMMR) endometrial carcinoma

DETAILED DESCRIPTION:
Phase II is a single-arm safety and efficacy study to explore the safety and initial efficacy of BAT1308 combined with platinum-containing chemotherapy. The first 6 patients (using 3+3 method) were included in the safe induction period, and 3 subjects were included first DLT assessment was performed. If there were less than 2 cases of DLT, 3 subjects were further included for DLT assessment Less than 2 cases of DLT in the total 6 cases were formally entered into the phase II study, if the phase II combination drug regimen was safe Phase II enrollment was stopped and phase III study was entered when the full treatment was controllable and the efficacy was in line with expectations. Phase I study is BAT1308 in combination with platinum-containing chemotherapy vs. placebo plus platinum-containing chemotherapy for advanced first-line treatment or A randomized, double-blind, multicenter clinical study of patients with recurrent dMMR endometrial cancer. PFS As the primary endpoint, optimal design. Stratified by the following random factors Histological randomization: according to disease status (stage III, IV, or relapse), prior pelvic extrinsic release Patients were stratified by treatment history (yes or no).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, female, voluntarily sign informed consent;
2. The patient must have one of the following types of endometrial cancer: a) Newly diagnosed stage III disease (lesions assessed as measurable according to RECIST 1.1 after surgery or diagnostic biopsy), b) newly diagnosed stage IV disease (small lesions assessed as measurable or unmeasurable according to RECIST 1.1 after surgery or diagnostic biopsy, and truly unmeasurable lesions need to be excluded, (such as ascites, pleural effusion, etc.) c) recurrent diseases (small foci assessed as measurable or unmeasurable according to RECIST 1.1, truly unmeasurable foci, such as ascites, pleural effusion, etc.),
3. There is little likelihood of cure with surgery/radiotherapy alone or in combination, or surgery or radiotherapy cannot be tolerated;
4. Have not received first-line systemic anticancer therapy. Prior chemotherapy is permissible only for patients with recurrent disease if it is received under adjuvant conditions (as part of prior/adjuvant anticancer therapy) and the interval between the last dose of chemotherapy and the date of subsequent recurrence is at least 6 months;
5. Subjects should meet the requirements of mismatch repair protein deficiency (dMMR) detected by the central laboratory of tumor specimen. Subjects should provide sufficient paraffin embedded (FFPE) specimens or sections (6 recommended, no less than 3) and be willing to undergo tumor tissue biopsies if needed for MMR status detection. The archived tissue must be a representative tumor specimen less than three years old, or an unstained continuous section of newly cut FFPE tumor tissue within six months, and the relevant pathological report of the above specimen must be provided. Fresh tissue specimens can be harvested by surgical excision and biopsy. Do not accept fine needle puncture and liquid based cytology (TCT) samples (i.e., samples that lack complete tissue structure and only provide cell suspension and/or cell smear); Decalcified bone metastatic tumor tissue specimens are not accepted;
6. Expected survival assessed by investigators ≥12 weeks;
7. The physical status score of the American Eastern Cancer Consortium (ECOG) is required to be 0 ~1 points;
8. Fertile female patients must have a negative serological pregnancy test within 7 days prior to the first dosing and be willing to use effective birth control/contraception to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Postmenopausal women must have amenorrhea for at least 12 months before they are considered infertile.

Exclusion Criteria:

1. Have endometrial leiomyosarcoma or other high-grade sarcoma, or endometrial stromal sarcoma.
2. Pregnant and lactating women;
3. Radical radiation therapy was received within 3 months before the first administration of the study drug. Note: Palliative radiotherapy for bone or superficial lesions is permitted, the course of treatment is according to local standards and has ended 14 days before the first dose. Radiotherapy that covers more than 30% of the bone marrow area within 28 days prior to initial dosing is not permitted; Received chemotherapy drugs for radiosensitization within 14 days prior to initial administration; Within 14 days prior to the first administration of the drug, have received the NMPA-approved Chinese patent medicine or treatment clearly with anti-tumor related functions, or the medical record clearly recorded in the anti-tumor purpose of Chinese herbal therapy;
4. are participating in the treatment stage of other clinical studies, or plan to start this study treatment less than 14 days from the end of drug treatment of the previous clinical study;
5. Have received live/attenuated vaccines and mRNA vaccines within 4 weeks prior to screening or plan to receive live/attenuated vaccines and mrna vaccines during the study period;
6. Previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.) or immunocostimulatory factors (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.) and other treatments targeting tumor immune mechanisms;
7. Before the first administration of antitumor therapy, there were still more than grade 1 aes (based on CTCAE v5.0) (except for alopecia, fatigue and other AE that could not be restored to grade 1 or less and would remain in a stable state for a long time as judged by researchers based on clinical conditions, and grade 2 peripheral neurotoxicity. Except for stable hypothyroidism after hormone replacement therapy); Those who had a history of ≥ grade 3 irAE or had discontinued immunotherapy for any grade of irAE;
8. Active pia meningeal disease or poorly controlled brain metastases. Patients with suspected or confirmed BMS were admitted if they were asymptomatic, had stable disease on imaging findings ≥28 days prior to first administration of the study drug, and did not require treatment (such as radiation therapy, surgery, or corticosteroid therapy) to control symptoms of BMS for 28 days prior to first administration of the study drug.
9. Patients who underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first use of the study drug, or who required elective surgery during the trial period;
10. Any active infection that requires systematic anti-infective therapy occurs within 14 days prior to the first administration of the investigational drug;
11. there are the following diseases infected: human immunodeficiency virus (HIV) infection; Active hepatitis B virus infection [hepatitis B surface antigen (HBsAg) positive, HBV deoxyribonucleic acid (HBV-DNA) test >500IU/ml or 103 copies /ml or greater than the upper limit of normal test unit]; HCV infection [HCV antibody and viral ribonucleic acid (HCV-RNA) test positive or greater than the upper limit of the normal value of the test unit]; Treponema pallidum antibody positive and RPR positive;
12. Subjects with untreated or under treatment for tuberculosis, including but not limited to tuberculosis; Patients who have received standardized anti-tuberculosis treatment and have been confirmed cured by the researchers can be included;
13. Known to have a history of severe allergy, or known subjects have had grade 3 or greater allergic reactions to macromolecular protein preparations/monoclonal antibodies or to any of the test drug components;
14. There is clinically significant hydronephrosis, which cannot be relieved by nephrostomy or ureteral stenting according to the investigators;
15. Subjects with uncontrolled pleural effusion, pericardial effusion, or abdominal effusion requiring repeated drainage;
16. Patients with active or prior autoimmune disease with a history of recurrence (excluding vitiligo, autoimmune thyroid disease that can be treated with hormone replacement therapy, type 1 diabetes);
17. Received systemic use of glucocorticoids (prednisone > 10mg/ day or equivalent dose of the same drug) or other immunosuppressants within 14 days prior to the first use of the study drug, except for the following: Treatment with topical, ocular, intraarticular, intranasal and inhaled glucocorticoids, and short-term prophylactic treatment with glucocorticoids (for example, to prevent hypersensitivity to contrast media);
18. Subjects with a history of noninfectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to initial administration;
19. have a history of serious cardiovascular and cerebrovascular disease, including but not limited to: ① New York Heart Association (NYHA) grade II or above heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) There are serious heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree Ⅱ-Ⅲ atrioventricular block, etc.; ③ Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first dose; (4) Clinically uncontrollable hypertension (defined in this protocol as systolic blood pressure > 160mmHg and/or diastolic blood pressure > 100mmHg despite antihypertensive therapy);
20. Uncontrolled/unstable thrombotic or hemorrhagic disease;
21. Patients with other active malignant tumors within 3 years prior to screening, except locally curable tumor species and those who have been cured;
22. Imaging examination showed that there were clear manifestations of tumor invasion of the thoracic great blood vessels
23. Subjects with a known history of psychotropic substance abuse or drug use that is thought to affect compliance with this study;
24. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
25. Subjects deemed unsuitable for participation in this study (considerations include but are not limited to: impact on compliance, safety and ethical considerations, impact on interpretation of study results, etc.).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
vital signs | Through study completion, 1 year
  Number of participants with abnormal vital signs
Physical examination | Through study completion, 1 year
  Number of participants with abnormal physical examination
Adverse events | From the first receipt of the investigational drug until 28 (+7) days after the last receipt of the investigational drug or the initiation of a new antitumor therapy, whichever occurs earlier，assessed up to 1 year
  Number of participants with various adverse events (AEs)
Clinical laboratory tests | Through study completion, 1 year
  Number of participants with abnormal clinical laboratory tests
Clinical auxiliary tests | Through study completion, 1 year
  Number of participants with abnormal clinical auxiliary tests
Dose-limiting toxicity (DLT) | From the first receipt of the investigational drug until 28 (+7) days after the last receipt of the investigational drug or the initiation of a new antitumor therapy，assessed up to 1 year
  DLT events and their incidence
Progression Free Survival | Tumor imaging assessments will be performed once every 6 (±7) days during the screening period, once every 6 (±7) days after initial dosing to 25 weeks, and once every 9 (±7) weeks，assessed up to 1 year，the screening period is 28 days
  Progression Free Survival（PFS ）in patients with advanced or recurrent dMMR endometrial cancer treated with BAT1308 combined with platinum-containing chemotherapy were compared with platinum-containing chemotherapy in first-line treatment by IRC according to RECIST V1.1.

SECONDARY OUTCOMES:
Initial efficacy | Tumor imaging assessments will be performed once every 6 (±7) days during the screening period, once every 6 (±7) days after initial dosing to 25 weeks, and once every 9 (±7) weeks，assessed up to 1 year
  Initial efficacy was assessed by investigators according to the solid tumor Efficacy Evaluation Criteria (RECIST V1.1)
Pharmacokinetic | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days(The first 12 subjects).
  Level of Cmax
Pharmacokinetic | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days(The first 12 subjects).
  Level of Tmax
Pharmacokinetic | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days(The first 12 subjects).
  Level of T1/2
Pharmacokinetic | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days(The first 12 subjects).
  Level of CL
Immunogenicity | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days
  Level of ADA
Immunogenicity | At the end of Cycel1Day1,cycle3Day1,Cycle5Day1,after Cycle5, for 9 weeks，assessed up to 1 year，each cycle is 28 days
  Level of NAb

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality, China